CLINICAL TRIAL: NCT06117644
Title: A Single-center, Prospective Study of the Efficacy of Double-dose Furmonertinib in the Treatment of Patients With Slow Osimertinib-resistant Non-small Cell Lung Cancer
Brief Title: The Efficacy of Double-dose Furmonertinib in the Treatment of Patients With Slow Osimertinib-resistant NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yong He, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: Posterior-coast
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation; Non Small Cell Lung Cancer Stage IIIA; Non-small Cell Lung Cancer Stage IV
Keywords: Non Small Cell Lung Cancer; EGFR Gene Mutation; Furmonertinib; Drug Resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Furmonertinib: The subjects will be treated with Furmonertinib (double dose, 160mg). The subjects were treated with drugs for 24 months until the tumor progressed (worsened) or died.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 40 mg/tablet, 4 tablets, QD

SUMMARY:
This study is a single-center, prospective, single-arm study of the efficacy of double-dose Furmonertinib in the treatment of patients with slow Osimertinib-resistant non-small cell lung cancer, mainly in patients with advanced non-small cell lung cancer with EGFR-sensitive mutations in stage IIIB or IV, slow drug resistance after treatment with Osimertinib, and no therapeutic target was found by secondary biopsy after drug resistance.

DETAILED DESCRIPTION:
According to the latest data released by the National Cancer Center in 2022, the incidence and mortality of cancer in China are increasing year by year. There are 4.064 million new cancer patients in China in 2016, with a total of 2.414 million cancer deaths. Among them, 824000 were new cases of lung cancer, accounting for 20.4%, and the number of lung cancer deaths was 657000, accounting for 27.2%. The morbidity and mortality of lung cancer ranked first among all malignant tumors. Non-small cell lung cancer (NSCLC) accounts for about 80% of all lung cancer types, of which epidermal factor growth receptor (EGFR) mutation is the most common driving gene for NSCLC. About 50% of Chinese patients carry this gene mutation. Exon 19 deletion mutation (19Del) and exon 21 L858R point mutation (L858R) are called "classical mutations", accounting for about 90% of all mutation types.

With the third generation of EGFR-TKI gradually entering the clinic, the survival benefits of patients with EGFR classical mutation positive NSCLC have been continuously broken through. FLAURA study showed that the median progression-free survival time (mPFS) of Osimertinib was significantly better than that of gefitinib in the first-line treatment of advanced NSCLC patients with positive EGFR mutation (18.9 months VS 10.2 months, HR 0.46 (P < 0.001). In addition, the third-generation domestic EGFR-TKI ametinib, vometenil and so on, have also been listed in China in recent years. No matter in terms of survival time or quality of life, the third generation of EGFR-TKI has brought clinically significant improvement to patients. At present, both foreign NCCN guidelines and domestic CSCO guidelines have taken the third generation of EGFR-TKI as the standard scheme for first-line treatment of EGFR classic mutation positive patients.

However, with the wide application of the third generation EGFR-TKI, the problem of drug resistance of the third generation TKI is becoming more and more obvious. The time of the third-generation TKI listing and application in China is concentrated around 2021, while the mPFS of the third-generation EGFR-TKI is concentrated between 18-22 months. Therefore, it can be expected that the problem of drug resistance in the third generation of TKI may continue to intensify in the next few years. At present, after the third generation-TKI resistance or progress, there is no standard and unified treatment plan. The third generation of TKI drug resistance has become a very urgent and huge clinical problem. Therefore, there is an urgent need to carry out clinical or real-world studies related to the third-generation TKI drug resistance to explore more or better solutions after the third-generation TKI drug resistance, so as to bring more potential treatment options for the third-generation TKI drug-resistant patients.

At present, the exploration direction of the third generation TKI drug resistance therapy includes immune combination therapy (such as Xindimazumab + chemotherapy + anti-angiogenic drugs), precision targeted combination therapy (EGFR-TKI combined with MET-TKI,EGFR-TK combined with RET-TKI, etc.), antibody coupling drugs (ADC), bispecific antibodies, fourth generation-EGFR-TKI and so on. However, the above treatments may face problems such as insufficient drug accessibility, excessive adverse reactions, or less than expected survival time. In addition to the above direction, after the third-generation-TKI resistance, the challenge of using the third-generation TKI with increased dose is also one of the options that may be used in clinical practice, which also shows preliminary clinical value in the real world.

Fumetinib methanesulfonate (AST2828) is the third generation irreversible TKI. At present, NMPA has approved fumetinib for first-line treatment of locally advanced or metastatic NSCLC patients with positive EGFR mutation (19Del/L858R), and second-line (posterior-line) treatment for patients with disease progression with T790M mutation during or after EGFR-TKI treatment. The results of its IIB phase clinical study showed that for advanced NSCLC patients with positive T790M mutation, the ORR at the recommended dose of 80mg/ days was as high as 74.1%, and the median PFS was 9.6 months. The results of III phase FURLONG study showed that the mPFS of advanced EGFR mutation positive (19Del/L858R) NSCLC patients treated withFurmonertinib was significantly better than that of gefitinib (20.8months VS 11.1months, HR=0.44,P < 0.0001). In general, the conventional dose of Furmonertinib showed a good therapeutic effect in both first-line and second-line treatment of advanced NSCLC with classical EGFR mutation.

At the same time, in phase I and I/II clinical trials, some patients received daily doses of 160mg (n = 53) and 240mg (n = 18), and no dose-limiting toxicity was observed. Compared with the 80mg dose group, the main increases in the incidence of adverse reactions were increased alanine aminotransferase (80mg 17.5% 1600240mg 35.2%), decreased white blood cell count (80mg 13.8% 1600240mg 29.6%), decreased neutrophil count (80mg 7.8% 1600240mg 18.3%), increased serum creatinine (80mg 7.5% 1600240mg 18.3), diarrhea (80mg 6.7% 1600240mg 15.5%). Anemia (80mg 6.0% metrology 1600240mg 23.9%). The main increased incidence of adverse reactions in the 160-240mg dose group compared with the 80mg dose group ≥ 3 was anemia (80mg 0% meme 1600240mg 4.2%). The results of this phase I/II study showed that increased doses of Furmonertinib maintained acceptable safety and tolerance.

Zheng et al reported a case of successful salvage treatment with Furmonertinib 160mg/d after Osimertinib resistance. The clinical efficacy of oxetinib in this patient lasted only 7 months, followed by sequential use of Furmonertinib160mg/d. After two weeks of treatment, the tumor was significantly reduced and the respiratory symptoms were significantly improved. At the same time, the intracranial lesions of the patients were completely relieved after 1 month of treatment. This case suggests that the use of increased doses of Furmonertinib may be a potential treatment option for patients with drug resistance to Osimertinib. Another real-world study explored the efficacy and safety of 160mg/d Furmonertinib in patients with three generations of EGFR-TKI drug resistance. In 39 patients, the median PFS and OS of Furmonertinib 160mg/d were 4.7 months and 7.53 months, respectively. Among them, it showed a better therapeutic effect for the third generation of TKI patients with intracranial progression, with a median PFS of 5.45months and a median OS of 9.75months. The main adverse reactions were anemia, lymphocytopenia, diarrhea and so on. No new safety signal was observed. This real-world study preliminarily validates the efficacy and safety of increased-doseFurmonertinib (160mg/d) in patients with third-generation TKI drug resistance.

To sum up, the researchers predict that a higher dose of 160mg/d in third-generation TKI-resistant patients may have a better benefit-risk ratio, which has the value of further exploration. Therefore, this real-world study intends to collect three generations of TKI-resistant patients who have been treated with increased doses of Furmonertinib. To further analyze the efficacy and safety of improving the dose of Furmonertinib in the third generation of patients with TKI drug resistance. To provide more evidence-based medical evidence for the treatment of the third generation of patients with drug resistance to TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. EGFRm NSCLC of local progression (IIIB stage) or metastasis (IV stage);
3. previously confirmed to have EGFR (Ex19del or L858R) mutation, or T790M, received Osimertinib treatment. According to Recist 1.1 imaging findings, the focus progressed slowly and there was no systemic explosive progress (definition of slow progress: disease control > 6 months, slightly increased tumor load and symptom score ≤ 1);
4. patients who intend to use Furmonertinib (double dose, 160mg) anticancer therapy;
5. At least one tumor lesion in the patient can meet the following requirements: it has not been irradiated in the past and can be accurately measured, the longest diameter of the baseline phase is ≥ 10mm (in the case of lymph nodes, short axis ≥ 15mm is required), and the measurement method can be chest CT or PET-CT, as long as repeated measurements can be completed accurately;
6. No treatable target was found in the second biopsy after drug resistance;
7. The survival time was more than 3 months;

Exclusion Criteria:

1. Patients who have been treated with Furmonertinib;
2. Patients who intend to use anticancer therapy other than Furmonertinib recently;
3. Contraindications for the use of Furmonertinib;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mainly targeted at IIIB or IV stage EGFR sensitive mutation advanced non-small cell lung cancer patients with slow drug resistance after Osimertinib treatment, and no treatable target was found by secondary biopsy after drug resistance.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Observation time 1-2 months.
  Objective response rate (ORR) including rate of CR and PR on based of RECIST 1.1

SECONDARY OUTCOMES:
OS | through study completion (36 months)
  Overall survival (OS) defined as the median time from randomization to death from any cause.
PFS | through study completion (36 months)
  Progression-free survival (PFS) the time from first dose of the study drug until the date of disease progression or death by any cause.
DCR | through study completion (36 months)
  Disease control rate (DCR) including rate of CR, PR and SD on based of RECIST 1.1
AE | through study completion (36 months)
  AE refers to any adverse medical event that occurs in patients who have taken a drug or in clinical research subjects, which is not necessarily causal to the drug.

IPD SHARING:
Plan to Share IPD: No